CLINICAL TRIAL: NCT01216553
Title: Home Oxygen Therapy in the Ambulatory Treatment of Bronchiolitis
Brief Title: Home Oxygen Therapy in Bronchiolitis
Acronym: O2-Rx
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: E. Michael Sarrell M.D, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 134/2010
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Infants; Nebulized Inhalation; RSV; Oxygen
MeSH Terms: conditions — Bronchiolitis | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypertonic inhalation + O2 (Active Comparator): oxygen for 30 minuets after inhalation of 3% saline 4 times daily
  Interventions: Other: Oxygen Therapy
- Epinephrine & bromhexine nebulized + O2 (Active Comparator): oxygen for 30 minuets after inhalation of racemic epinephrine with bromhexine 4 times daily
  Interventions: Other: Oxygen Therapy

INTERVENTIONS:
Other: Oxygen Therapy — 1 lt/min oxygen via nasal cannulae intermittently for 30 minuets 4 times daily for 7 days
  Other Names: O2

SUMMARY:
The aim of the study was to investigate the utility and safety of home management of home oxygen therapy in acute bronchiolitis. A matched case-control study, of one hundred and thirty five infants aged less than 12 months diagnosed bronchiolitis with hypoxia attending a pediatric community clinic will be randomly assigned to receive oxygen with or without standard nebulized therapy. Nebulized treatment with either 0.1% epinephrine diluted in bromhexine, or 3% hypertonic saline. Intermittent oxygen treatment will be administered 6 times daily for 7 days. Primary outcome measures will be emergency department visits/hospitalization secondary outcome measures will be changes in Bronchiolitis Caregiver Diary Score.

DETAILED DESCRIPTION:
Bronchiolitis is an infection of the bronchiolar epithelium. It is associated with profound submucosal and adventitial edema, increased secretion of mucus, and obstructed flow in the small airways, leading to hyperinflation, atelectasis, and wheezing. Respiratory syncytial virus (RSV) is responsible for the majority of cases .Bronchiolitis is the most frequent lower respiratory tract infection with high morbidity, and the leading cause of hospitalization in young children. Studies from developed countries report an incidence hospitalization of 30 per 1000 children in the first year of life and an annual mortality rate of 1.82-2 per 100,000 live births. The cost of treatment is about $2.5 billion yearly. One group from the United States estimated the annual hospital costs for bronchiolitis at $365-$691 million.

Of children who develop bronchiolitis during the first 2 year of life, approximately 1 in 10 ( 3% of all infants in the USA) will be hospitalized furthermore, a substantial proportion of infants remain in the hospital to receive oxygen until their hypoxia has improved.

The current in hospital treatment for acute viral bronchiolitis is mainly supportive, consisting of supplemental oxygen, suction and hydration . Airway edema and sloughing of respiratory epithelia cell cause mismatching of ventilation and perfusion and subsequently reduction in oxygenation (PaO2 and Spo2). Emergency Department referral (ED) and Hospital admission (HA) admission, have increased secondary to increase sensitivity of pulse oximetry for detection of hypoxia ( compared with clinical observation. The therapeutic role of bronchodilators although of questionable clinical importance is commonly used A recent review reported has shown short-term improvement in clinical scores, but no improvement in oxygenation or rate of hospitalization. Neither systemic glucocorticoids nor antibiotics appear to have any clinically significant effect on the disease course. Antiviral agents (Ribavirin) are indicated only in children with a serious underlying disorder. Trials with chest physiotherapy using vibration and percussion techniques failed to reduce the severity of the illness, length of hospitalization, or oxygen requirements, and treatment with nebulized furosemide ,inhaled interferon alpha-2a (Roferon A) ,and rhDNase proved ineffective.

Clinicians are now influenced significantly in their decision for Emergency Department referral and hospitalization of patient with respiratory disease. We hypothesized that adding short term home intermittent oxygen therapy for 7 days to other treatment modalities will reduce hypoxias and Emergency Ward referral. The aim of the present study was to compare the outcome of this combined treatment with oxygen with other medical modalities to oxygen alone and with placebo in children with RSV bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Infants, aged less than 24 months treated for acute viral bronchiolitis in a pediatric ambulatory clinic in central Israel, during the winter season (December through April) of 2011-2013. The clinical diagnosis will be based on findings of a first clinical bronchiolitis requiring oxygen for hypoxia.

Exclusion Criteria:

* Infants with chronic diseases, such cardiorespiratory disease, cystic fibrosis or neonatal asthma, malignancy or immunodeficiency will be excluded, as will be infants in severe distress (respiratory rate >80breaths/min, heart rate >200beats/min, BCD score >13, SpO2). Infants who had recovered from chronic neonatal lung disease of prematurity will be included. In addition, we will excluded infants who had received corticosteroids or bronchodilators in any form within 14 days before presentation and infants whose parents refused to participate or were unable to complete the Bronchiolitis Caregiver Diary Score.

Ages: 8 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-05 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Home oxygen therapy in the ambulatory treatment of bronchiolitis | 1 month
  Primary outcome measures of the study will be the number of emergency room visits or hospitalizations within two weeks of enrollment in the study.

SECONDARY OUTCOMES:
Home oxygen therapy in the ambulatory treatment of bronchiolitis | 1 month
  Secondary outcome measures the change in bronchiolitis caregiver diary (BCD) score.
daycare(patients) and work (parents) lost because of the illness. | 1 month
  Number of day that patient has missed from daycare, forcing one parent to miss work

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Gani- Hdar Clinic, Petah Tikva
  - Clalit health services -Gani Hadar Clinic, Tel Aviv